CLINICAL TRIAL: NCT06544031
Title: Increasing the Level of Knowledge and Reflecting on Attitudes With the "Healthy Nutrition" Training to the Individuals in the Nursing Home in Izmir Buca Social Life Campus
Brief Title: Enhancing Knowledge and Attitudes Through the 'Healthy Nutrition' Education Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Democracy University (Other)
Responsible Party: Principal Investigator, Aysel Başer, Asistant Prof., Izmir Democracy University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: NutEdu1
Record Dates: First submitted 2024-07-22; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Health Behavior; Nutrition, Healthy; Educational Activities
Keywords: Solomon Four Group Experimental Design; Healthy Nutrition Attitude Scale,; Nutrition Knowledge Level,; Healthy Nutrition Education,; Geriatrics,; Healthy Nutrition
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Intervention Model Description: The study employs a Solomon Four Group Design, which includes parallel groups for evaluating the impact of the "Healthy Nutrition" education program on nutritional knowledge and attitudes among elderly individuals.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental Education-Pre and Post Test G1 and G2 (Experimental): Arm Title: Experimental Pre-education Group 1-2 Arm Type: Experimental Description: Participants receive a pre-test, followed by the educational intervention, and then a post-test.
  Intervention(s): Healthy Nutrition Education
  Interventions: Behavioral: Healthy Nutrition Education Program
- Control Group with only Pre and Post test G3 and G4 (No Intervention): Arm Title: Control Group 1 Arm Type: No Intervention Description: Participants receive a pre-test and a post-test without any intervention.
- Experimental Education- Post Test G5 (Experimental): Arm Title: Experimental Group 2 Arm Type: Experimental Description: Participants receive the educational intervention followed by a post-test.
  Intervention(s): Healthy Nutrition Education
  Interventions: Behavioral: Healthy Nutrition Education Program
- Control Group with only Post test G6 (No Intervention): Arm Title: Control Group 2 Arm Type: No Intervention Description: Participants receive only a post-test without any intervention.

INTERVENTIONS:
Behavioral: Healthy Nutrition Education Program — The program consists of two sessions totaling 2 hours. The first session includes a traditional presentation on healthy nutrition, and the second session involves an interactive question and answer segment. The intervention aims to improve nutritional knowledge and attitudes towards healthy eating among elderly residents.
  Arms: Experimental Education- Post Test G5; Experimental Education-Pre and Post Test G1 and G2

SUMMARY:
This study aims to assess the impact of a "Healthy Nutrition" education program on the knowledge and attitudes towards healthy eating among elderly individuals residing in a Social Life Campus. The study utilizes a Solomon four-group experimental design, involving participants divided into an experimental group and a control group. Participants were selected based on their ability to effectively participate in the education program, with no psychological or neurological illnesses

DETAILED DESCRIPTION:
The study was conducted using an experimental method to examine the effect of healthy nutrition education on the nutritional awareness and attitudes of older adults residing in a social living home for the elderly (SLHO) within the Izmir Buca Social Life Campus. The study was conducted between 01 February 2023 and 01 June 2024.

The study was conducted among elderly residents aged 60 years and older, without psychiatric or neurological diseases. Participants were divided into experimental and control groups. The Solomon Four Group Design was utilized to compare the effects of the intervention, including pretest and posttest measurements to account for time-dependent changes.

Ethical approval for the study was obtained from the Izmir Democracy University Non-Interventional Clinical Research Ethics Committee, with the decision numbered 2023/02-13, dated 01/02/2023. All participants signed an informed consent form before the study commenced.

The "Healthy Nutrition" education program included two sessions lasting a total of 2 hours. The first session involved traditional presentation-based education, while the second session was an interactive question and answer session. Only the experimental group received this training.

Data collection involved:

Sociodemographic Data Form: Collected basic demographic information such as age, gender, and educational status.

Nutrition Knowledge Scale (NKS) and Healthy Nutrition Attitude Scale (HNAS): Used to measure participants' nutritional knowledge levels and attitudes. These scales were administered both before and after the educational intervention to assess the potential impact of the program.

ELIGIBILITY:
Inclusion Criteria:

* Must be a resident at İzmir Buca Social Life Campus.
* Must be willing to participate voluntarily.
* Must not have any psychological or neurological disorders (e.g., dementia, Alzheimer's disease) that would prevent participation in the training.

Exclusion Criteria:

* Non-voluntary participation: Individuals who are not willing to participate voluntarily.
* Presence of psychological or neurological disorders (e.g., dementia, Alzheimer's disease) that would prevent participation in the training.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2023-07-15 (Actual); Primary Completion 2023-08-03 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Change in Nutrition Knowledge | Pre-test (baseline) and post-test (immediately after the intervention for experimental groups; same time points for control groups).
  The change in nutrition knowledge levels before and after the intervention will be assessed using the Nutrition Knowledge Scale (NKS). Developed by Yılmaz et al. in 2021, the NKS evaluates adult nutrition knowledge across food and nutrient knowledge, food preparation and cooking methods, and the relationship between nutrition and health. The scale includes both positive and reverse-scored items, rated on a 5-point Likert scale. The total score ranges from 0 to 126, with higher scores indicating greater nutrition knowledge. Specific cut-off points are as follows: <79 for low knowledge, 79-89 for medium, 90-100 for high, and >101 for very high knowledge levels.
  Ref: Öngün Yılmaz, H., et al. (2021). Nutrition Knowledge Scale (NKS): Development, factor structure, and validation for healthy adults. Progress in Nutrition, 23(3). Available at: Mattioli 1885 Journals.

SECONDARY OUTCOMES:
Change in Healthy Nutrition Attitudes | Pre-test (baseline) and post-test (immediately after the intervention for experimental groups; same time points for control groups).
  The change in attitudes towards healthy nutrition before and after the intervention will be evaluated using the Healthy Nutrition Attitude Scale (HNAS).
  Measurement Tool: The Healthy Nutrition Attitude Scale (HNAS) was developed by Demir and Cicioğlu in 2019. It consists of 21 items categorized into four factors: Nutrition Knowledge (NK), Emotional Attitude towards Nutrition (EAN), Positive Nutrition (PN), and Poor Nutrition (PN). The scale is rated on a 5-point Likert scale, with higher scores indicating a more favorable attitude toward healthy nutrition.
  Scoring: The possible score ranges are:
  21 points: Very low attitude 23-42 points: Low attitude 43-63 points: Moderate attitude 64-84 points: High attitude 85-110 points: Ideal level of healthy nutrition attitude

CONTACTS AND LOCATIONS:
Overall Officials: Aysel Baser, Study Director — Izmir Democracy University
Locations (1):
- İzmir Democracy University, Izmir, Konak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data (IPD) that will be shared includes de-identified data on demographics, pre-test and post-test scores, and responses to the Nutrition Knowledge Scale (NKS) and Healthy Nutrition Attitude Scale (HNAS). Data will be shared upon request for research purposes and will be available from [12.2024] to [12.2029]. Researchers can request access by contacting the principal investigator at [aysel.akpinar@gmail.com].
Supporting Information: SAP
Time Frame: The data will be available starting six months after the study results are published and will remain available for five years.
Access Criteria: Data will be shared with anyone who requests it via email. The reason for this access period is to allow sufficient time for secondary analyses, replication studies, and to contribute to the broader scientific community. Researchers who wish to access the data should send a request to the provided email address.

REFERENCES:
- [Derived] Yetkin B, Baser A. Enhancing knowledge and attitudes through the 'healthy nutrition' education program: a Solomon four-group experimental study with older adults at a social life campus. BMC Geriatr. 2025 Jul 2;25(1):436. doi: 10.1186/s12877-025-05861-5. PMID 40604505
- See also: Attitude Scale for Healthy Nutrition (ASHN): Validity and Reliability Study — http://dergipark.org.tr/tr/pub/gaunjss/issue/45377/559462
- See also: Nutrition Knowledge Scale (NKS) — http://www.mattioli1885journals.com/index.php/progressinnutrition/article/view/11030